CLINICAL TRIAL: NCT00627185
Title: Dental Tobacco Control.Net:Improving Practice
Acronym: DTC
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X030814016; R01DA017971 (NIH)
Record Dates: First submitted 2008-02-14; First posted 2008-02-29 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2010-08

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco control; Tobacco cessation; Tobacco use
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation; Tobacco Use | interventions — Patient Portals; Quality Assurance, Health Care; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention group (dental practices) that received the interactive motivational website for patient tobacco cessation
  Interventions: Behavioral: Internet-delivered continuing professional development
- 2 (Placebo Comparator): Control group (dental practices) that did not receive any materials or resources on tobacco cessation. This is a wait-list control.
  Interventions: Other: No intervention arm

INTERVENTIONS:
Behavioral: Internet-delivered continuing professional development — Interactive motivational website for dentists and hygienists with practice improvement resources, discussion forum, and educational cases on cessation counseling with email reminders.
  Other Names: Internet; Quality Assurance, Health Care; Tobacco Use Cessation
  Arms: 1
Other: No intervention arm
  Arms: 2

SUMMARY:
This is a randomized, controlled trial (RCT) to test the efficacy of an internet continuing dental education intervention designed to increase tobacco cessation counseling in dental practices. The intervention involves surveying practices regarding preventive care, surveying adult patients about their tobacco habits and preventive care provided by dental practice and training/educating the dentist and office staff on tobacco cessation. With patients who smoke and indicate that they have quit, we followed up with testing their saliva for the presence of cotinine. We have enrolled general dentists and periodontists who practice in the Southeastern United States.

DETAILED DESCRIPTION:
Tobacco use has been described as the number one behavioral health problem of our time with a projected 8.4 million total smoking related deaths worldwide by the year 2020. Current clinical practice guidelines entitled "Treating Tobacco Use and Dependence" provide a summary of evidence-based recommendations. Despite the evidence of tobacco risk and the efficacy of tobacco control interventions, 30% of current smokers report that they have never been advised to stop smoking by a healthcare provider. Nearly half (47.9%) of dentists report they have never intervened to assist tobacco users in quitting. Our intervention is designed to improve the rate of tobacco cessation advice delivered in dental practices.

This proposal is in response to the request for applications "Translational Research in Dental Practice-based Tobacco Control Interventions" (RFA: DE-03-007). Our exploration of barriers and facilitators will assist in clarifying processes that influence translation of tobacco-related knowledge into clinical dental practice. Our trial will integrate theoretically grounded methods of provider behavior change, medical informatics, and tobacco control research to translate guidelines into dental clinical practice. We will avoid a "one-size-fits-all" approach by tailoring strategies for tobacco cessation counseling to individual practices. The intervention will be longitudinal, with updates and continuous access for dentists and dental staff over 2 years. Our evaluation will extend from processes of care to patient outcomes. Ancillary analyses will assess differences in tobacco counseling rates associated with practice, provider, and patient-level variables including disparities in counseling by race. To assess the relative impact of various components of the multi-modal intervention, we will conduct secondary analyses of the association of amount of use of each specific component with frequency of tobacco cessation counseling within the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* general dental practices that have internet access
* Periodontal practices that have internet access
* patients of participating dental or periodontal practices

Exclusion Criteria:

* patients who were 18 years of age and younger

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2003-09; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Our primary outcome measures are patient-reported provider delivered tobacco screening and tobacco cessation advice. | Baseline, 8-months post-intervention, and 24-months post-intervention

SECONDARY OUTCOMES:
Point prevalence smoking cessation | six-months after index visit for patients who smoke

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Houston, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Houston TK, Funkhouser E, Allison JJ, Levine DA, Williams OD, Kiefe CI. Multiple measures of provider participation in Internet delivered interventions. Stud Health Technol Inform. 2007;129(Pt 2):1401-5. PMID 17911944
- [Result] Houston TK, Richman JS, Ray MN, Allison JJ, Gilbert GH, Shewchuk RM, Kohler CL, Kiefe CI; DPBRN Collaborative Group. Internet delivered support for tobacco control in dental practice: randomized controlled trial. J Med Internet Res. 2008 Nov 4;10(5):e38. doi: 10.2196/jmir.1095. PMID 18984559
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- [Derived] Houston TK, Delaughter KL, Ray MN, Gilbert GH, Allison JJ, Kiefe CI, Volkman JE; National Dental PBRN Collaborative Group. Cluster-randomized trial of a web-assisted tobacco quality improvement intervention of subsequent patient tobacco product use: a National Dental PBRN study. BMC Oral Health. 2013 Feb 23;13:13. doi: 10.1186/1472-6831-13-13. PMID 23438090